CLINICAL TRIAL: NCT04501692
Title: Endotracheal Tube-mounted Camera Assisted Intubation Versus Videolaryngoscopic Intubation in Patients With Expected Difficult Airway - a Prospective Randomized Trial
Brief Title: VivaSight-SL Versus Videolaryngoscopy in Expected Difficult Airway
Acronym: VivaOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VivaOP
Record Dates: First submitted 2020-08-02; First posted 2020-08-06 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Airway Management

STUDY DESIGN:
Intervention Model Description: randomized 1:1
Who Masked: Participant
Masking Description: device for intubation may not be blinded for provider or investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VivaSight (Experimental): Intubated with a VivaSight-SL endotracheal tube.
  Interventions: Procedure: VivaSight
- Conventional (Active Comparator): Intubated by videolaryngoscopy.
  Interventions: Procedure: Videolaryngoscopy

INTERVENTIONS:
Procedure: VivaSight — see above
  Arms: VivaSight
Procedure: Videolaryngoscopy — see above
  Other Names: comparator
  Arms: Conventional

SUMMARY:
Patients requiring endotracheal intubation for elective surgery with an expected difficult airway are randomized to be intubated either by a) videolaryngoscopy or b) an endotracheal tube-mounted camera.

DETAILED DESCRIPTION:
Endotracheal intubation is required for different surgical procedures for mechanical ventilation and to prevent aspiration of secretions. Endotracheal intubation is usually performed by direct laryngoscopy (DL), but this technique may fail in patients with a difficult airway, i.e. during otorhinolaryngologic or oral and maxillofacial surgery. Besides fiberoptic intubation that is regarded as gold standard, videolaryngoscopy (VL) has evolved as a valuable alternative technique in patients with a difficult airway. However, VL has its limitations and may also fail due to insufficient visualization of the larynx. An endotracheal tube with an integrated camera (VST, VivaSight-SL, Ambu A/S, Ballerup, Denmark) may allow for direct guidance of the tube and may aid in endotracheal intubation in difficult airway patients. This tube has been evaluated in intensive care patients and in patients with morbid adiposity compared to DL, but there is a paucity of data in difficult airway patients, so far.

Therefore, we aim to test the VST in difficult airway patients compared to VL in a prospective randomized non-inferiority trial.

Patients will be assessed for eligibility in the Anesthesiology Pre-assessment Clinic of the University Medical Center Hamburg-Eppendorf prior to elective surgery.

All patients receive a structured preoperative airway assessment in accordance with standard operating procedure of the Department of Anesthesiology, University Medical Center Hamburg-Eppendorf using the implemented in-house algorithm for the prediction of difficult airway management and the Simplified Airway Risk Index (SARI).

Patients randomized to the intervention group will be intubated with a VST. Depending on gender and patient's size, tubes with inner diameters of 7.0, 7.5, and 8.0 are available. The tubes camera is connected to an Ambu aView monitor (Ambu A/S, Ballerup, Denmark). Patients randomized to the control group are intubated with a C-MAC videolaryngoscope (Karl Storz SE & Co. KG, Tuttlingen, Germany) with a Macintosh type blade size 3 or 4 blade.

Anesthesia management, the choice of the blade and tube size, as well as the use of adjuncts like stylets, introducers or forceps or airway optimization maneuvers (e.g. backward upward rightward pressure [BURP] and optimum external laryngeal manipulation [OELM]) will be left to the discretion of the attending physician.

All intubations are recorded through the monitors for later review (e.g. Cormack-Lehane and POGO-score).

Based on an expected endtidal fraction of oxygen after intubation of 80% with a standard deviation of 8%, and a noninferiority margin of 10%, 2x 24 patients are required with errors of α=0.025 and β=0.2 (PASS version 08.0.6, NCSS, LLC. Kaysville, UT, USA).

All participating physicians are anesthesiology residents or fellows. To avoid a bias that may occur due to different skills for VL compared to the VST, physicians participating in this study take part in a structured manikin airway training. The age and months of work experience of the participating anesthetists will be assessed within a questionnaire. It has been shown that novice physicians are able to reliably intubate a manikin with the VST after a 30 min training session of DL and VST. For VL, it has been shown that novice physicians may intubate manikins set up to a difficult airway scenario after a brief introduction and five intubations with the VL and that anesthesiology residents may quickly adopt the use of the C-MAC VL.

Therefore, participating physicians are trained for 30 min under the supervision of an independent anesthetist before participating in this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring general anesthesia with transoral tracheal intubation for elective surgery
* Age ≥ 18
* Preoperative airway assessment reveals an expected difficult airway (rated by the responsible anesthetist in the Pre-assessment Clinic based on the existing in-house algorithm)

Exclusion Criteria:

* Pregnant or breastfeeding woman
* Confirmed indications for awake fiberoptic intubation especially due to enoral, pharyngeal tumors, abscesses or other processes
* Planned endotracheal intubation without deep anesthesia or neuromuscular blocking agents (e.g. awake videolaryngoscopy)
* Required transnasal tracheal intubation (e.g. for surgical reasons)
* Requirement of special endotracheal tubes such as laser or RAE tubes for surgical reasons
* Patients at risk for pulmonary aspiration who qualify for rapid sequence induction
* Loose teeth
* Denial of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-08-27 (Actual); Primary Completion 2021-02-12 (Actual); Study Completion 2021-02-12 (Actual)

PRIMARY OUTCOMES:
first-pass success | 15 minutes
  percentage of successful intubations with one attempt
end-tidal oxygen fraction | 15 minutes
  the lowest end-tidal oxygen fraction within two minutes after successful intubation after a standardized preoxygenation

SECONDARY OUTCOMES:
overall success rate | 15 minutes
  percentage of successful intubations with the allocated procedure
time to successful intubation | 15 minutes
  time until an endotracheal airway access is established
time to successful intubation with one attempt | 15 minutes
  time until an endotracheal airway access is established in patients that are intubated at first attempt
intubation difficulty | 15 minutes
  subjective rating on a visual analogue scale of the difficulty of airway management and questionnaire
end-tidal carbondioxide fraction | 15 minutes
  the highest end-tidal carbondioxide fraction within two minutes after successful intubation
number of attempts | 15 minutes
  total number of attempts until airway established
aspiration | 15 minutes
  percentage of patients that vomit and aspirate during intubation
esophageal intubation | 15 minutes
  percentage of accidental esophageal intubation attempts
hypoxia | 15 minutes
  percentage of patients with a desaturation below a pulsoximetric saturation of 80%
hypotension | 15 minutes
  percentage of patients with a systolic blood pressure below 70 mmHg
intubating conditions | 15 minutes
  grades according to Cormack-Lehane and POGO

CONTACTS AND LOCATIONS:
Overall Officials: Joern Grensemann, MD, Study Chair — Universitätsklinikum Hamburg-Eppendorf; Martin Petzoldt, MD, Study Chair — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- Universitätsklinikum Hamburg-Eppendorf, Hamburg, Hamburg, Germany